CLINICAL TRIAL: NCT06128928
Title: REDES: a Peer Network and mHealth Community Health Worker (CHW) Model to Improve COVID-19 Vaccination Among Latinos
Brief Title: Connecting Friends and Health Workers to Boost COVID-19 Vaccination in Latino Communities
Acronym: REDES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00345930; R01MD017364 (NIH)
Record Dates: First submitted 2023-11-10; First posted 2023-11-13 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: COVID-19; Vaccine
Keywords: COVID-19 vaccine uptake; Latino; vaccine hesitancy; Network referrals
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REDES: Motivational interviewing training (Experimental): Participants in this arm will receive training on motivational interviewing (MI) to promote vaccine acceptance and uptake with their networks. The training will be led by community health workers on how to use MI to address vaccine hesitancy using a guiding approach, open-ended questions, affirmations, reflections, and summaries.
  Interventions: Behavioral: REDES
- Control: COVID-19 vaccine information (Active Comparator): Participants in the control condition will receive a brief community health worker-led training about the safety and efficacy of the vaccine. Participants will have the opportunity to ask clarifying questions from the community health workers during the training.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: REDES — Training on motivational interviewing (MI) led by community health workers on how to use MI to address vaccine hesitancy using a guiding approach, open-ended questions, affirmations, reflections, and summaries.
  Arms: REDES: Motivational interviewing training
Behavioral: Control — Brief CHW-led training about the safety and efficacy of the COVID-19 vaccine. Participants will have the opportunity to ask clarifying questions from the CHWs during the training.
  Arms: Control: COVID-19 vaccine information

SUMMARY:
The goal of this clinical trial is to find out which approach works better in getting more of the friends and connections of Latino adults get vaccinated against COVID-19.

The main questions this study aims to answer are:

1. Can teaching people to use motivational interviewing help more friends and connections of Latino adults get the COVID-19 vaccine compared to just giving information about the vaccine?
2. What are the things that make it easier or harder for Latinos and networks to get the COVID-19 vaccine?
3. How does this intervention work in practice so that it can be made available to more people in the future

The researchers will compare the vaccine rates of the friends and connections of Latinos who have been trained in motivational interviewing with those who have only been given information about the COVID-19 vaccine. This will help figure out which method works best to encourage more people to get vaccinated.

DETAILED DESCRIPTION:
This study will test the efficacy of an intervention REDES ("Networks") - a social network intervention - to address COVID-19 vaccine hesitancy and uptake among a cohort of Latinos and networks. 300 index participants who have taken the COVID-19 vaccine will be recruited. Half of the index participants (n=150) will be randomized to the experimental group and will receive training on motivational interviewing to promote vaccine acceptance and uptake with networks. Index participants in the control group (n=150) will receive updated information about the COVID-19 vaccine. In addition, unvaccinated primary and secondary network members of indexes will be recruited for study participation and COVID-19 vaccination. All participants will be followed prospectively at 6, 12, and 18 months after baseline intake. The specific aims are: 1) Evaluate the efficacy of the REDES intervention to promote COVID-19 vaccine uptake among Latinos; 2) Examine ongoing barriers and facilitators of vaccine uptake among Latinos and networks to tailor the intervention and address new challenges, and 3) Evaluate the implementation determinants and outcomes of REDES to inform future broad-scale implementation.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for index participants (eligibility for index participants is intended to select participants who are less vaccine hesitant):

* Age 18 years or older, and
* Self-identifies as Hispanic/Latino, and
* Living in Maryland, and
* Has received at least one COVID-19 vaccine/booster in the last 12 months.

Eligibility criteria for primary and secondary network members (peers):

Eligibility for peers is intended to select for participants who are more vaccine hesitant (e.g. unvaccinated, or have not received at least one COVID-19 vaccine/booster in the last 12 months)

* 18 years old or older, and
* Self-identifies as Hispanic/Latino, and
* Living in Maryland, and
* Provide a study coupon to verify that they were referred by an index or a primary network member, and
* Has not received at least one COVID-19 vaccine/booster in the last 12 months.

Exclusion Criteria:

* Previously participated in the study
* Lacks capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-07-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccine status among networks | Up to 18 months
  Number of network participants who receive the COVID-19 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Page, MD, Principal Investigator — Johns Hopkins University; Cui Yang, PhD, Principal Investigator — Rutgers University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States